CLINICAL TRIAL: NCT01051128
Title: Continuous Intrathecal Baclofen Infusion for the Management of Chronic Spasticity
Brief Title: Continuous Intrathecal Baclofen Infusion for Chronic Spasticity
Acronym: CIBI
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was never started. Full IDE-approval not obtained. new IDE will be submitted
Sponsor: Flowonix Medical (Industry)
Responsible Party: Janelle Arrambide, Medasys, Incorporated
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G090276
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Spasticity
Keywords: neurological disorders; multiple sclerosis; stroke; cerebral palsy; spinal cord; brain injuries; neurodegenerative diseases
MeSH Terms: conditions — Muscle Spasticity; Nervous System Diseases; Multiple Sclerosis; Stroke; Cerebral Palsy; Brain Injuries; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spasticity. Baclofen (Experimental): This study is a non-randomized, open-label, multi-center study of the Prometra Programmable Implantable Pump System in the administration of Lioresal® intrathecal (baclofen) in patients suffering from severe muscle spasticity of spinal origin.
  Interventions: Device: Prometra Programmable Implantable Pump System

INTERVENTIONS:
Device: Prometra Programmable Implantable Pump System — The Prometra Programmable Pump is a battery-operated, implantable, programmable infusion pump that dispenses drug solution into the intrathecal space through an implanted infusion catheter. All functions of the system (e.g., dosing) are controlled externally using a hand-held, battery-operated programmer.

SUMMARY:
The purpose of this clinical investigation is to demonstrate product performance of the Prometra Programmable Pump System in the delivery of intrathecal Lioresal® (baclofen) for the management of severe spasticity.

DETAILED DESCRIPTION:
The Prometra Programmable Pump is a battery-operated, implantable, programmable infusion pump that dispenses drug solution into the intrathecal space through an implanted infusion catheter. All functions of the system (e.g., dosing) are controlled externally using a hand-held, battery-operated programmer. Lioresal Intrathecal (baclofen) is indicated for use in the management of severe spasticity. Spasticity is a major problem that has long challenged traditional medical treatment. While the incidence of spasticity is not known with certainty, it likely affects over half a million people in the United States and over 12 million worldwide. Spasticity is associated with some very common neurological disorders such as: multiple sclerosis, stroke, cerebral palsy, spinal cord and brain injuries. Chronic spasticity seriously restricts normal daily activities and reduces the quality of life for many patients.

ELIGIBILITY:
Inclusion Criteria:

The overall goal of this study is to choose patients most likely to experience therapeutic success while reducing the likelihood of risks, complications and adverse events.

Patients meeting all of the following criteria will be eligible for enrollment in the study:

1. Patient with a history of severe chronic spastic hypertonia in the lower extremities lasting at least 6 months who:

   * fail to respond to maximum recommended doses of antispasmodic medications including baclofen, or
   * those who experience intolerable CNS side effects at effective oral doses
2. Patient is >21 years of age
3. Patient, or legally authorized representative (LAR), has provided written informed consent to participate in the study
4. Investigator considers the patient willing and able to fulfill all study requirements
5. Investigator has documented attempts to eliminate factors that can contribute to an increase in spasticity (e.g. infection)
6. Patient has had a successful trial of Lioresal® for the management of the target spasticity.

Exclusion Criteria:

Patients meeting any of the following criteria are to be excluded from the study:

1. Patient has MRI of the spine documenting structural abnormality preventing adequate CSF flow. (If the patient has a medical condition that contraindicates screening MRI, the investigator should proceed with the closest appropriate study i.e. CT scan, X-ray, to rule out any spinal abnormalities that would prevent intrathecal drug administration.)
2. Patient's anatomy is not large enough to accommodate the pump's size and weight.
3. Patient has a systemic infection.
4. Patient has renal insufficiency as evidenced by a baseline serum creatinine of >2.0 mg/dl.
5. Patient has a history of a bleeding disorder.
6. Patient has a history of blood clots such as deep vein thrombosis (DVT) or pulmonary embolism (PE) within 1 year of enrollment.
7. Patient is pregnant or breast-feeding, or is of child-bearing potential and not employing effective birth control.
8. Patient has known allergies or sensitivities to pump system materials (e.g., silicone rubber, titanium, polyphenylsulfone, acetal resin, polyvinylidene fluoride, tungsten).
9. Patient has known allergies to Lioresal® (baclofen), or would be contraindicated for Lioresal® based on the drug labeling.
10. Patient has other implantable electronic cardiac devices (i.e. pacemaker, defibrillator, CRT system)
11. Patient has an occupation where he/she would be exposed to high current industrial equipment, powerful magnets or transmitting towers, such as, electricians, electrical engineers or MRI technicians.
12. Patient is participating in another clinical trial.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is: A change in the average lower extremity spasticity score as measured by the Modified Ashworth Scale | 3 months

SECONDARY OUTCOMES:
Secondary Endpoints include: Change in overall spasm frequency as measured by the Penn Spasm Frequency Scale. Change in overall Quality of Life as measured by the SF 36 and PSQI. SAE-free survival. DRAE-free survival. Tabulation of device complications. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Levy, MD, PhD, Principal Investigator — Northwestern University Hospital